CLINICAL TRIAL: NCT00003196
Title: Induction of Mixed Hematopoietic Chimerism in Older Patients With B-Cell Malignancies and in Selected Other Diseases, Using Low Dose TBI , PBSC Infusion and Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil to be Followed by Donor Lymphocyte Infusion: A Pilot Study.
Brief Title: Low-Dose Total Body Irradiation and Donor Peripheral Blood Stem Cell Transplant Followed by Donor Lymphocyte Infusion in Treating Patients With Non-Hodgkin Lymphoma, Chronic Lymphocytic Leukemia, or Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1225.00; NCI-2012-00592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); #1225.00A; 1225.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage II Multiple Myeloma; Stage III Multiple Myeloma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Drug Therapy; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (irradiation, transplant, immunosuppression, DLI) (Experimental): CYTOREDUCTION: If necessary, patients with advanced malignancies undergo cytoreductive chemotherapy to reduce tumor size at discretion of primary physician and study investigators.
  CONDITIONING REGIMEN: Patients undergo low-dose total-body irradiation followed by allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine IV BID on days -1 to 0 and then PO BID on days 1-35 with taper to day 56. Patients also receive mycophenolate mofetil PO BID on days 0-27.
  POST-TRANSPLANT DLI: Patients with mixed chimerism on day 56 and no evidence of GVHD undergo DLI over 30 minutes on day 65 and may receive up to 3 additional infusions in the absence of GVHD and disease progression or persistence. Patients who have not achieved mixed chimerism at day 56 undergo DLI if complete response is not obtained after a 2 month monitoring period.
  Interventions: Drug: chemotherapy; Radiation: total-body irradiation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Biological: therapeutic allogeneic lymphocytes

INTERVENTIONS:
Drug: chemotherapy — Undergo cytoreductive chemotherapy
  Other Names: chemo
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSC transplant
Biological: therapeutic allogeneic lymphocytes — Undergo DLI
  Other Names: ALLOLYMPH

SUMMARY:
This pilot clinical trial studies low-dose total body irradiation and donor peripheral blood stem cell transplant followed by donor lymphocyte infusion in treatment patients with non-Hodgkin lymphoma, chronic lymphocytic leukemia, or multiple myeloma. Giving total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them. Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether mixed hematopoietic chimerism can be safely established using a non-myeloablative conditioning regimen in patients with non-Hodgkin lymphoma (NHL), chronic lymphocytic leukemia (CLL) and multiple myeloma.

II. To determine whether mixed chimerism, established with non- myeloablative conditioning regimens, can be safely converted to full donor hematopoietic chimerism by infusions of donor lymphocytes (DLI).

OUTLINE:

CYTOREDUCTION: If necessary, patients with advanced malignancies undergo cytoreductive chemotherapy to reduce tumor size at discretion of primary physician and study investigators.

CONDITIONING REGIMEN: Patients undergo low-dose total-body irradiation followed by allogeneic peripheral blood stem cell (PBSC) transplant on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine intravenously (IV) twice daily (BID) on days -1 to 0 and then orally (PO) BID on days 1-35 with taper to day 56. Patients also receive mycophenolate mofetil PO BID on days 0-27.

POST-TRANSPLANT DLI: Patients with mixed chimerism on day 56 and no evidence of graft-vs-host disease (GVHD) undergo DLI over 30 minutes on day 65 and may receive up to 3 additional infusions in the absence of GVHD and disease progression or persistence. Patients who have not achieved mixed chimerism at day 56 undergo DLI if complete response is not obtained after a 2 month monitoring period.

After completion of study treatment, patients are followed up at 4, 6, 12, 18, and 24 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 49 years and < 66 years with NHL, CLL and multiple myeloma who are not eligible for autologous transplantation or have failed prior autologous transplantation; patients with NHL and CLL must have failed prior therapy with an alkylating agent and/or fludarabine; patients with multiple myeloma must have stage II or III disease and received prior chemotherapy
* Patients < 50 years of age with NHL, CLL and multiple myeloma at high risk of regimen related toxicity through prior autologous transplant or through pre-existing chronic disease affecting kidneys, liver, lungs, and heart will be considered on a case by case basis and presented to professional clinical counselor (PCC)
* Patients < 66 years of age with other diseases treatable by allogeneic bone marrow transplant (BMT) whom through pre-existing chronic disease affecting kidneys, liver, lungs, and heart are considered to be at high risk for regimen related toxicity using standard high dose regimens; autografting must also be contraindicated in these patients and they must be approved for this protocol by both PCC and by the principal investigator; the following diseases are the likely candidates but other less common diseases may be considered and approved by PCC:

  * Myelodysplastic syndromes
  * Myeloproliferative syndromes
  * Acute leukemia in remission
  * Chronic myelogenous leukemia (CML) in 2nd chronic phase
  * Hodgkin's disease
* Selected patients with any of the above diagnosis who are (a) older than 65 years and < 75 years with a Karnofsky score >= 70 and who, apart from age, fulfill eligibility criteria, or (b) < 66 years but ineligible solely because of renal dysfunction; these patients must be approved for transplant by both PCC and the principal investigator
* DONOR: Human leukocyte antigen (HLA) genotypically identical sibling
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)
* DONOR: Age < 75

Exclusion Criteria:

* Eligible for autologous transplantation
* Patients with rapidly progressive high grade NHL
* History of central nervous system (CNS) involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Patients with a creatinine clearance < 50 ml/min
* Cardiac ejection fraction < 40% or cardiac failure requiring therapy
* Severe defects in pulmonary function testing (defects are currently categorized as mild, moderate and severe) as defined by the pulmonary consultant, or receiving supplementary continuous oxygen
* Total bilirubin > 2 x the upper limit of normal
* Serum glutamate pyruvate transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) 4 x the upper limit of normal
* Karnofsky score < 50
* Patients with poorly controlled hypertension
* DONOR: Identical twin
* DONOR: Age less than 12 years
* DONOR: Pregnancy
* DONOR: Infection with human immunodeficiency virus (HIV)
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness
* DONOR: Failure to meet Fred Hutchinson Cancer Research Center (FHCRC) criteria for donation as described in the Standard Practice Guidelines

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 1997-09 (Actual); Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Incidence of GVHD, myelosuppression, and infections | Up to 5 years
  At the conclusion of the study, all unexpected toxicities will be summarized and reported.
Greater than 10% incidence of treatment-related mortality (TRM) after PBSC infusion, defined as death without evidence of disease progression | Within 65 days of transplant
Greater than 20% incidence of TRM after DLI, defined as death without evidence of disease progression | Within 12 months of DLI
Proportion of patients who successfully achieve mixed chimerism | Up to 5 years
  The proportion of patients who successfully establish mixed chimerism in each group (patients with NHL, CLL or multiple myeloma vs patients with other malignancies) will be estimated and corresponding confidence intervals will be presented.
Proportion of patients with mixed chimerism who successfully achieve full donor chimerism | Up to 5 years
  The proportion of patients with mixed chimerism who are successfully converted to full donor chimerism in each group (patients with NHL, CLL or multiple myeloma vs patients with other malignancies) will be estimated and corresponding confidence intervals will be presented.

SECONDARY OUTCOMES:
Response of malignancy to DLI | Up to 5 years
  Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.
Incidence of myelosuppression after initial PBSC transplant | Up to day 56
  Defined as (absolute neutrophil count [ANC] < 500 for > 2 days, platelets < 20,000 for > 2 days). Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.
Incidence of aplasia after DLI | Up to day 90
  Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.
Incidence of grades 2-4 acute GVHD after DLI | Up to day 90 post-DLI
  Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.
Incidence of grades 2-4 acute GVHD after PBSC infusion | Up to day 56
  Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.
Incidence of chronic extensive GVHD after DLI | Up to 1 year post-DLI
  Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.
Dose of cluster of differentiation (CD)3+ cells required to convert mixed to full lymphoid chimeras | Up to 5 years
  Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.
Incidence of non-relapse mortality | Up to 5 years
  Examined separately in the two groups of patients, and reported in a descriptive manner with confidence intervals presented.

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (5):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
- Universitaet Leipzig, Leipzig, Germany
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241